CLINICAL TRIAL: NCT02106338
Title: Randomized, Double-blind, Placebo-controlled, Multiple Ascending Dose Phase I Trial to Determine the Safety and Pharmacokinetics of CRS3123 Administered Orally to Healthy Adults
Brief Title: Phase I Trial to Determine the Safety and Pharmacokinetics of CRS3123.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 10-0009; HHSN272201500007I
Record Dates: First submitted 2014-03-13; First posted 2014-04-08 (Estimated); Last update posted 2016-06-13 (Estimated); Status verified 2014-09

CONDITIONS: Clostridium Difficile Infection
Keywords: follow-up to 10-0008, Clostridium difficile, dose-escalating, CRS3123
MeSH Terms: conditions — Clostridium Infections | interventions — REP 3123

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (3):
- Cohort A (Experimental): 10 subjects (8 active, 2 placebo) receive a single oral dose of 200 mg CRS3123 or placebo every 12 hours for 10 days
  Interventions: Other: Placebo; Drug: CRS3123
- Cohort B (Experimental): 10 subjects (8 active, 2 placebo) receive a single oral dose of 100 or 400 mg CRS3123 or placebo every 12 hours for 10 days
  Interventions: Other: Placebo; Drug: CRS3123
- Cohort C (Experimental): 10 subjects (8 active, 2 placebo) receive a single oral dose of 600 mg CRS3123 or placebo every 12 hours for 10 days
  Interventions: Other: Placebo; Drug: CRS3123

INTERVENTIONS:
Other: Placebo — Placebo capsules have the same inert components as CRS3123; 2 subjects randomized in each cohorts recieve 200mg, 400mg; and 600mg, or 100mg are planned respectively given orally every 12 hours for 10 days
Drug: CRS3123 — CRS3123, a methionyl-tRNA synthetase inhibitor, formulated in 100 and 200 mg capsules; 8 subjects randomized in Cohorts A through C receive doses of 200 mg, 400 mg; and 600 mg or 100mg are planned respectively given orally every 12 hours for 10 days.

SUMMARY:
This is a Phase I, single center, randomized, placebo-controlled, double-blind, multiple ascending dose study to evaluate the safety and tolerability of CRS3123, a methionyl-tRNA synthetase inhibitor. In this study, doses of 200, 400, and 600 mg, or 100mg are planned and will be given orally every 12 hours for 10 days. Up to 30 healthy male and female subjects 18 to 45 years, inclusive. The primary objective: of the study is to determine the safety and tolerability of escalating doses of CRS3123 following oral administration of multiple doses to healthy adults. The study duration is 46 weeks.

DETAILED DESCRIPTION:
This is a Phase I, single center, randomized, placebo-controlled, double-blind, multiple ascending dose study to evaluate the safety and tolerability of CRS3123,a fully synthetic, oral, antimicrobial that targets methionyl-tRNA synthetase of gram-positive bacteria, including Clostridium difficile. This protocol will study oral doses of 200, 400, and 600 mg, or 100mg given orally every 12 hours for 10 days. Subjects will be divided into 3 cohorts, A, B, and C. Cohorts A and C will be given 200mg and 600mg of CRS3123 or placebo.The dose for cohort B and study progression and dose escalation to Cohorts B and C will require a full (planned) SMC review of all safety data obtained through Day 18. Should safety data review of the 200 mg dose result in an unfavorable safety profile, the study design allows for reduction in dose to 100 mg to be given in Cohort B. If this is the case, there will be no Cohort C. Up to 30 healthy male and female subjects 18 to 45 years, inclusive. The primary objective: of the study is to determine the safety and tolerability of escalating doses of CRS3123 following oral administration of multiple doses to healthy adults. The secondary objective will be to determine the plasma, urine and fecal concentrations and systemic exposure of CRS3123 after multiple oral doses.The study duration is 46 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Men and women 18 to 45 years of age, inclusive
* Ability to understand the consent process and study procedures
* Informed consent obtained and signed
* Subjects agree to be available for all study visits. Subjects will be asked if they have any travel plans, and whether staff could use alternate contact information that will be provided.
* General good health, without current medical illness or clinically significant abnormal physical examination findings that classify the subject as other than healthy as determined by study investigators
* Negative serum pregnancy test at screening on the day of admittance to the inpatient phase I unit for all female subjects
* Negative alcohol screen per phase I unit standard procedures (Breathalyzer) and urine toxicology screen for barbiturates, benzodiazepines, THC, cocaine, opiates, methamphetamines, TCA, methadone, MDMA (ecstasy), oxycodone, and amphetamines on screening and the day of admission to the inpatient phase.
* Agrees not to consume any alcohol 48 hours prior to admission or outpatient study visits.
* Body mass index (BMI) of < 35 [weight (kg)]/[height (m)^2]
* Agreement by subjects with reproductive potential to use an adequate method of contraception during the study and for 4 weeks after the initiation of study drug administration. Female subjects must agree to the use of TWO reliable methods of contraception starting on screening day, while receiving study drug and for 4 weeks after the initiation of study drug administration, which can include: condoms, spermicidal gel, diaphragm, hormonal or non-hormonal intrauterine device, oral contraceptive pill, and depot progesterone injections. If a male subject is sexually active, the subject and his partner will each use at least one of the listed contraceptive methods. Women who have had a surgical sterilization procedure (tubal ligation, oophorectomy, or hysterectomy) are not required to use another birth control method
* Potential subjects must be willing to adhere to the following prohibitions and restrictions during the course of the study to be eligible for participation: - Strenuous exercise (e.g., long distance running > 5km/day, weight lifting, or any physical activity to which the subject is not accustomed) is to be avoided while confined to the Clinical Unit and for at least 72 hours prior to initial study drug administration and the scheduled follow-up visits Day 18 and 29.

Exclusion Criteria:

* Medical condition that precludes participation, including the following:

  * Hypertension with confirmed systolic blood pressure >140 mmHg or confirmed diastolic blood pressure >90 mmHg, measured with vital signs after 10 - 15 minutes of rest. Abnormal measures may be repeated twice more (for a total of 3 times) at 5-10 minute intervals
  * Current diagnosis of pulmonary disease
  * Current diagnosis of asthma, which has required use of asthma medications within the past year
  * History of or current diagnosis of diabetes mellitus
  * Autoimmune disorder, such as lupus, Wegener's, rheumatoid arthritis
  * History of malignancy except low-grade skin cancer, (i.e., basal cell carcinoma, which has been surgically cured)
  * Chronic renal, hepatic, or pulmonary disease or gastrointestinal tract condition that could interfere with the absorption of the study drug (e.g., surgical resection of significant proportions of the stomach or bowel, gastric bypass, gastric banding, irritable bowel syndrome, inflammatory bowel disease)
  * History of known Clostridium difficile infection
  * History of cardiac rhythm abnormality including Wolff-Parkinson-White syndrome
  * History of prolonged QT interval
  * History of ovarian cysts
* Prolongation of QTcF interval (>450msec). Clinically significant abnormal electrocardiogram at screening in the judgment of the investigator, or based on the formal ECG reading by a Cardiologist; history of any cardiac abnormalities, including conduction abnormalities such as Wolff-Parkinson-White, dysrhythmias, or coronary artery disease
* Laboratory values outside the expanded ranges in Appendix B for the following tests: Blood Cell Counts (white blood cell counts [WBC], with differential hemoglobin, platelets), Serum Chemistry (sodium, potassium, chloride, CO2, calcium, glucose, creatinine, BUN, CK, AST, ALT, AP, total bilirubin, protein, albumin, amylase, lipase), and Urinalysis (dipstick for glucose, protein and blood, and microscopic urinalysis if dipstick is abnormal and with provisons for re-testing in menstruating females in Section 7.16). If CK is above normal range at baseline, but not clinically significant, the subject can be included.
* Positive serology results for HIV, HBsAg, and HCV antibodies
* Febrile illness with temperature documented >38 degrees C within 7 days of dosing
* Pregnancy or breastfeeding
* Known allergic reactions to study drug components, including ingredients present in the formulation.
* Treatment with another investigational drug within 30 days of dosing
* Lack of ability to fully understand the informed consent. This will be determined and documented, per Phase I Unit procedures, by the recruiter/interviewer assigned Phase 1 Unit personnel after explaining the consent and observing the subject reading the consent.
* Ingestion of prescription medications, grapefruit juice, or St John's Wort starting 14 days before dosing. Women may use oral contraceptives.
* Ingestion of herbal supplements or over-the-counter medications starting 7 days before dosing
* Use of any form of tobacco, including cigarette smoking, pipe smoking, or oral tobacco; if a former smoker or tobacco user, the subject must not have used tobacco for 30 days before screening based on reported medical history
* Any specific condition that, in the judgment of the Investigator, precludes participation because it could affect subject safety
* Subjects may not have donated blood in the 8 weeks prior to study entry and agree to not donate blood during and for 6 weeks following their active participation in the study.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Estimated)
Dates: Start 2014-06; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
The sequential review of reported adverse events | Up to Day 29
The changes from baseline in key ECG findings | Up to Day 29
The changes from baseline in vital sign measurements | Up to Day 29
The changes from baseline in findings on physical examination. | Up to Day 29
The changes from baseline of hematology test | Up to Day 29
The changes from baseline of urinalysis test | Up to Day 29
The changes from baseline of clinical chemistry test | Up to Day 29

SECONDARY OUTCOMES:
Urine CRS3123 concentrations at multiple specified time points following dose administration. | Day 2, 4, 6, 8, 10-12
Fecal CRS3123 concentrations before oral administration of CRS3123 | Day -1
Plasma CRS3123 concentrations at multiple specified time points following dose administration. | Day 2, 4, 6, 8, 10-12
Fecal CRS3123 concentrations at multiple specified time points following dose administration | Day 2, 4, 6, 8, 10-12
Urine CRS3123 concentrations before oral administration of CRS3123 | Day -1
Plasma CRS3123 concentrations before oral administration of CRS3123 | Day -1

CONTACTS AND LOCATIONS:
Locations (1):
- Quintiles Phase I Services - Overland Park, Overland Park, Kansas, United States

REFERENCES:
- [Derived] Lomeli BK, Galbraith H, Schettler J, Saviolakis GA, El-Amin W, Osborn B, Ravel J, Hazleton K, Lozupone CA, Evans RJ, Bell SJ, Ochsner UA, Jarvis TC, Baqar S, Janjic N. Multiple-Ascending-Dose Phase 1 Clinical Study of the Safety, Tolerability, and Pharmacokinetics of CRS3123, a Narrow-Spectrum Agent with Minimal Disruption of Normal Gut Microbiota. Antimicrob Agents Chemother. 2019 Dec 20;64(1):e01395-19. doi: 10.1128/AAC.01395-19. Print 2019 Dec 20. PMID 31685472